CLINICAL TRIAL: NCT05362331
Title: Feasibility of a "Companion for CAR-T" Web App During Chimeric Antigen Receptor T-cell Therapy
Brief Title: Companion for CAR-T Web App During Chimeric Antigen Receptor T-cell Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Contract issues
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 212527; NCI-2022-03845 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-01

CONDITIONS: Lymphoma; Leukemia; Plasma Cell Dyscrasia
Keywords: Web Application; CAR-T Therapy
MeSH Terms: conditions — Lymphoma; Leukemia; Paraproteinemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Companion for CAR-T Web Application (CC) (Experimental): Enrolled participants and caregivers will receive access to the CC web application during the participants Chimeric Antigen Receptor T-cell (CAR-T) therapy. Key components include (1) educational videos and materials, (2) appointment calendars and 'Appointment Companion' features to prepare for clinical appointments, and (3) tools to assist with vital sign and neurological monitoring at home.
  Interventions: Other: Web Application

INTERVENTIONS:
Other: Web Application — Internet based application
  Other Names: Companion for CAR-T Web Application; CAR-T Web Application (CC); CAR-T Web App

SUMMARY:
The complex logistics and unique toxicities of chimeric antigen receptor T-cell (CAR-T) therapy require intensive patient education and careful monitoring. The Companion for CAR-T (CC) web app may be able to assist with patient education and preparation, communication between patients and their multidisciplinary teams, and home-based toxicity monitoring.

DETAILED DESCRIPTION:
This is a single-arm pilot study assessing the feasibility and acceptability of the Companion for CAR-T (CC) web app among patients receiving commercially available CAR-T therapies.

Primary Objectives:

I. To evaluate the feasibility of the CC web app. II. To evaluate the acceptability of the CC web app to patients.

Secondary Objectives:

I. To quantify the incidence of fevers being reported via the CC web app. II. To quantify the incidence of electronic Immune Effector Cell-Associated Encephalopathy (eICE) deficits being recorded via the CC web app.

Exploratory Objectives:

I. To explore patient perceptions regarding the CC web app. II. To explore usage patterns regarding the CC web app. III. To explore trends in patient-reported quality of life (QOL), values, and stressors over time during CAR-T therapy.

IV. To explore responses to abnormal findings reported or recorded using the CC web app

Participants will be given access to the web application from beginning at the day of study enrollment through Day +100 following CAR-T therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a hematologic malignancy (including any plasma cell dyscrasia, any type of lymphoma, or any type of leukemia).
* Planned receipt of an FDA-approved CAR-T therapy at University of California, San Francisco (UCSF) as standard of care.
* Patient proficiency in spoken and written English.
* Caregiver proficiency in spoken and written English.
* Age >= 18 years old

Exclusion Criteria:

* FDA-approved CAR-T therapy being administered as part of a prospective industry-sponsored trial, for example registrational trials of CAR-T therapy versus salvage chemotherapy or CAR-T therapy as an off-label line of therapy.

  *However, patients who receive an FDA-approved CAR-T therapy through an Expanded Access Program for non-conforming products (or any observational, non-interventional analysis of CAR-T products) are eligible.
* Lack of ownership of a personal computing device, tablet device, or smartphone.
* Refusal of patient and/or caregiver to sign up for a UCSF MyChart account.

  *Participants and caregivers who do not have a MyChart account at enrollment but are willing to create one will receive assistance from the study team to do so.
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could - in the opinion of the study's Principal Investigator (PI) - interfere with provision of informed consent or compliance with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who access all four CC web application modules at least once | Up to 6 months
  The percentage of participants who access all four CC web application modules at least once from the date of study enrollment through Day +100 after CAR-T therapy will be reported. To meet the acceptability criteria, a threshold of 70% of participant engagement or higher must be met.
Percentage of participants agreeing or strongly agreeing with helpfulness of CC web application. | 1 day
  Percentage of participants agreeing or strongly agreeing with the statement, "The Companion for CAR-T web app was helpful during my experience with CAR-T therapy." from a one time assessment administered between Day +29 and Day +100 following CAR-T therapy will be reported. This question ranks the helpfulness of the CC application on a scale of 1 (strongly disagree) to 5 (strongly agree). Participants must select an item score of 4 (agree) or 5 (strongly agree). To meet the feasibility criteria, a threshold of 70% of participant agreement or higher must be met.

SECONDARY OUTCOMES:
Number of times that temperature >= 38. degrees Celsius (°C) is reported | Up to 26 days
  The number of times (pooled across all patients) that an internal body temperature >= 38.0°C is reported by the participants via the CC web application between Day +2 to Day +28 following CAR-T therapy.
Number of times an Electronic immune effector-cell associated encephalopathy assessment (eICE) is reported | Up to 26 days
  The number of times (pooled across all patients) that a new eICE deficit is recorded via the CC web application between Day +2 to Day +28 following CAR-T therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Banerjee, MD, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No